CLINICAL TRIAL: NCT06372470
Title: Personalised Dose Optimisation of Zestril Supported by the Digital Blood Pressure Diary in a Primary Care Environment in England: Pragmatic Observational Pilot Study for Remote Hypertension Treatment
Acronym: OptiZest
Status: Completed | Type: Observational
Sponsor: Closed Loop Medicine (Industry)
Collaborators: Pharmanovia (Industry)
Responsible Party: Sponsor
Other Study IDs: CLM-HTN-005
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Uncomplicated Hypertension
MeSH Terms: interventions — Lisinopril

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Arm: Single cohort
  Interventions: Other: Zestril

INTERVENTIONS:
Other: Zestril — N/A, this is an observational study.

SUMMARY:
A pragmatic observational proof-of-concept study which aims to determine the feasibility of a remote titration clinic, assisted by home blood pressure monitoring and digital solutions, and assess its impact on real-world outcomes. By incorporating home blood pressure monitoring, the study seeks to offer a promising solution for personalised drug titration and self-management, potentially enhancing patient outcomes while optimising Zestril utilisation

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older.
2. Patients diagnosed with uncomplicated essential (primary) hypertension eligible for Zestril per SmPC for hypertension management.
3. Participants must provide written informed consent to participate in the study, including agreeing to adhere to the study procedures.
4. Have access to and be able to use a suitable smartphone independently, running either iOS version 15 or later or Android version 10 or later.

Exclusion Criteria:

1. Clinically significant abnormal blood results as judged by the investigator (exclude patients with known renal impairment).
2. History of clinically important medical conditions that would compromise a patient's ability to participate safely (including an allergic reaction to Zestril/lisinopril or any other medicine and/or other contraindications and interactions listed in Zestril's SmPC).
3. Patients with a strongly activated renin-angiotensin-aldosterone system (in particular, renovascular hypertension, salt and /or volume depletion, cardiac decompensation, or severe hypertension) as per SmPC
4. Participants who are unwilling or unable to participate in remote study procedures, including home BP monitoring, remote consultations, and data submission as judged by the investigator.
5. Any condition associated with poor compliance including alcoholism or drug dependence.
6. Participants with cognitive impairments or language barriers that hinder their ability to understand and comply with study instructions and e-questionnaires.
7. Failure to satisfy the investigator of fitness to participate for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Uncomplicated primary hypertension cohort in England
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-18 (Actual)

PRIMARY OUTCOMES:
Achieving target Home Blood Pressure | 12 weeks
  The number and percentage of patients achieving target Home Blood Pressure (Home Systolic Blood Pressure [HSBP] less than 135 and Home Diastolic Blood Pressure [HDBP] less than 85 mmHg for adults aged under 80; below 145/85 mmHg for adults aged 80 and over) at the optimal dose of Zestril at Week 12.

SECONDARY OUTCOMES:
Reduction in systolic blood pressure (SBP) | 12 weeks
  Mean change in SBP from baseline to the end of study Week 12
Reduction in diastolic blood pressure (DBP) | 12 weeks
  Mean change in DBP from baseline to the end of study Week 12
The time to achieve BP Control (BPC) | 12 weeks
  Median time from baseline to first achieving HBP control
Patient daily adherence to prescribed medication | 12 weeks
  Participants' daily adherence to Zestril, assessed using the digital diary, with adherence success defined as adherence to prescribed medication on 80% or more days during the 12-week titration period
Adherence to collecting data using the electronic BP diary | 12 weeks
  Adherence to collecting data using a digital diary will be determined by the percentage of the titration period during which patients input data into the blood pressure digital diary. Success will be defined as achieving 80% or more data input
Patients' thoughts and feelings about BP/treatment | 12 weeks
  Patient's thoughts and emotions about BP/Treatment assessed using the Brief Illness Perception Questionnaire (B-IPQ)
Discontinuation of Zestril due to unwanted side effects | 12 weeks
  Number and percentage of patients discontinuing Zestril due to unwanted side effects assessed at Week 12 using data collected from medical notes and withdrawal forms
Number and type of spontaneously reported unwanted side effects | 12 weeks
  Number and type of spontaneously reported unwanted side effects, assessed at Week 12 using data reported during each consultation (Week 2,4,6,8,10,12)
User experience and feasibility of the blood pressure digital diary | 12 weeks
  User experience and feasibility of the blood pressure digital diary assessed at Week 12 using the User Experience Questionnaire (UEQ)

CONTACTS AND LOCATIONS:
Overall Officials: Serge Engamba, Principal Investigator — Lead Principal Investigator
Locations (1):
- Norwich Health Centre, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: No